CLINICAL TRIAL: NCT03871621
Title: The Echocardiographic Left Ventricular Functional Changes of Uncontrolled Diabetes by the Intervention of Dapagliflozin Treatment Trial (ELUCIDATE)
Brief Title: Left Ventricular Functional Changes of Uncontrolled Diabetes by Dapagliflozin Treatment Trial
Acronym: ELUCIDATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18MMHIS149e
Record Dates: First submitted 2019-01-26; First posted 2019-03-12 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Cardiac remodeling; SGLT2 inhibitor; T2DM; Dapagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Hypoglycemic Agents; Metformin; Sulfonylurea Compounds; meglitinide; Thiazolidinediones; Insulin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin add-on group (Active Comparator): T2D subjects aged 20-80 years, presenting with HbA1C 7.1-9.0%, preserved kidney function (defined as estimated glomerular filtration rate (eGFR) > 60 mL/min/1.73 m2), preserved LV function (defined as EF ≥ 50% by echocardiographic screening in the initial 2-week run-in period), and those treated with oral anti-diabetic drugs (except SGLT2i) and/or insulin therapy at least 3 months prior to the study were randomised to Dapagliflozin (10 mg/qd) add-on group.
  Interventions: Drug: Diabetes Medicines; Drug: Dapagliflozin
- Standard of care (SOC) group (Active Comparator): T2D subjects aged 20-80 years, presenting with HbA1C 7.1-9.0%, preserved kidney function (defined as estimated glomerular filtration rate (eGFR) > 60 mL/min/1.73 m2), preserved LV function (defined as EF ≥ 50% by echocardiographic screening in the initial 2-week run-in period), and those treated with oral anti-diabetic drugs (except SGLT2i) and/or insulin therapy at least 3 months prior to the study were randomised to SOC treatment group.
  Interventions: Drug: Diabetes Medicines

INTERVENTIONS:
Drug: Diabetes Medicines — Anti-diabetic medications except SGLT2 inhibitors
  Other Names: Metformin; Sulfonylureas; Meglitinides; Thiazolidinediones; α-glucosidase inhibitor; Inhibitors of dipeptidyl peptidase 4; Insulin
Drug: Dapagliflozin — Dapagliflozin tablet (10 mg)
  Other Names: Farxiga
  Arms: Dapagliflozin add-on group

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of the SGLT2 inhibitor dapagliflozin, as compared with standard care of diabetes, on left ventricular (LV) structural and functional change in asymptomatic type 2 diabetes mellitus (DM) patient.

DETAILED DESCRIPTION:
The ELUCIDATE trial is a prospective, open label, randomized, active-controlled 'proof of concept'single centre study conducted in Mackay Memorial Hospital, Taipei, Taiwan. It is designed to clarify the LV remodeling by using Speckle-Tracking echocardiography to measure cardiac global longitudinal strain (GLS).

A cohort of 90 type 2 DM patients with normal LV ejection fraction will be randomized to either dapagliflozin 10 mg/die or to standard of care group as an active comparator. The study consists of 5 visits (see Table 1) and will last half an year, which has been ongoing since February 2019.

The primary outcomes are to detect the changes in LV mass index and cardiac GLS from baseline to 6 months after treatment initiation. The secondary outcomes include changes from baseline to 6 months in anthropometric measures, atrial-ventricular mechanics measurements, HbA1C,Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), epicardial fat and plasma biomarkers regarding cardiomyocyte remodeling and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female affected by type 2 diabetes mellitus (T2D) for at least 6 months.
* Age ≥ 20 and ≤ 80 years.
* HbA1c levels 7.1%~9.0% .
* On stable (at least 3 months) antidiabetic therapy with SGLT2 inhibitors naive.
* On stable (at least 3 months) cardio-active therapies (e.g. anti-hypertensive drugs, diuretics or drugs for hyperlipidemia).
* Preserved kidney function as defined by estimated glomerular filtration rate(eGFR)> 60 mL/min/1.73m2.
* Preserved left ventricular function defined as EF ≥ 50% by echocardiographic screening.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

* Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site).
* Previous enrolment or randomisation in the present study.
* Participation in another clinical study with an investigational product during the last 3 months.

The exclusion criteria that follow are for example only; include, exclude, modify or add other criteria as appropriate.

* Refuse or inability to give informed consent.
* Patients unlikely to comply with the protocol or unable to understand the nature and possible consequences of the study.
* Employees of the investigator or study centre (i.e. principal investigator, sub-investigator, study coordinators, other study staff, employees, or contractors of each), with direct involvement in the proposed study or other studies under the direction of that investigator and/or study centre, as well as family members of the employees or the investigator.
* Pregnancy or active breast feeding.
* History of hospitalization for heart failure.
* History of stage C or D heart failure.
* History of myocardial infarction.
* History of cardiac dysrhythmia.
* Patients with a known hypersensitivity to Dapagliflozin or any of the excipients of the product.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Cardiac global longitudinal strain (GLS) | Baseline to Week 24
  The primary outcome is to measure the change in cardiac GLS from baseline to 6 months after dapagliflozin treatment compared to standard diabetes care.
Left ventricular mass index | Baseline to Week 24
  The primary outcome is to measure the change in LVMi from baseline to 6 months

SECONDARY OUTCOMES:
Anthropometric measures by body mass index (BMI) | Baseline to Week 24
  Body weight in kilograms, body height in meters Body weight and height will be combined to report BMI in kg/m^2 Compare the change in anthropometric measures from baseline to 6 months
Blood pressure | Baseline to Week 24
  Change in SBP/DBP level (mmHg) over 24 weeks
HbA1c | Baseline to Week 24
  Change in HbA1c (%) by echocardiographic measurement over 24 weeks
Fasting glucose | Baseline to Week 24
  Change in fasting glucose level over 24 weeks
Homeostatic Model Assessment of Insulin Resistance, HOMA-IR | Baseline to Week 24
  Change in HOMA-IR over 24 weeks
Plasma biomarker: N-terminal pro-brain natriuretic peptide (NTproBNP) | Baseline to Week 24
  Change of NT-proBNP level (pg/mL) over 24 weeks
transforming growth factor beta 1 (TGF-β1) | Baseline to Week 24
  Change of TGF-β1 level (μg/L) over 24 weeks
Plasma biomarker: Growth differentiation factor-15 (GDF-15) | Baseline to Week 24
  Change of GDF-15 level (ng/L) over 24 weeks
tumor necrosis factor receptor I (TNF-RI) | Baseline to Week 24
  Change of TNF-RI level (ng/mL) over 24 weeks
Plasma biomarker: fatty acid binding protein 4 (FABP-4) | Baseline to Week 24
  Change of FABP-4 level (IU/mL) over 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No individual participant data share plan

REFERENCES:
- [Derived] Lin JL, Liu SC, Liu TF, Chuang SM, Huang CT, Chen YJ, Lee CC, Chien MN, Hou CJ, Yeh HI, Chiang CE, Hung CL. ELUCIDATE Trial: A Single-Center Randomized Controlled Study. J Am Heart Assoc. 2024 May 7;13(9):e033832. doi: 10.1161/JAHA.123.033832. Epub 2024 Apr 19. PMID 38639353